CLINICAL TRIAL: NCT06263348
Title: A Multicenter Post-Marketing Observational Study to Evaluate the Long-Term Safety of Dorzagliatin in Patients With Type 2 Diabetes Mellitus
Brief Title: A Post-Marketing Safety Study of Dorzagliatin in Patients With Type 2 Diabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Collaborators: Shanghai Branch, KunTuo Medical Research and Development (Beijing) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMM0601
Record Dates: First submitted 2024-02-05; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Type2diabetes
Keywords: Post-Marketing; long term Safety; Dorzagliatin
MeSH Terms: interventions — Dorzagliatin

STUDY DESIGN:
Intervention Model Description: The marketed product - Dorzagliatin tablet (HuaTangNing®) is used as the study drug. During this study, the dosage and administration of Dorzagliatin tablets will be completely in accordance with the investigator's judgment based on the package insert and the patient's condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dorzagliatin group (Experimental): Dorzagliatin tablet (75 mg, BID) treatment for 52 weeks
  Interventions: Drug: Dorzagliatin tablets

INTERVENTIONS:
Drug: Dorzagliatin tablets — During the study, patients should follow the dosing instructions from the investigator, which are made according to the package insert and the patients' conditions.

SUMMARY:
The primary objective of this study is to evaluate the long-term safety of Dorzagliatin in a larger population of type 2 diabetes mellitus patients by collecting the post-marketing clinical safety data of Dorzagliatin.

DETAILED DESCRIPTION:
This study adopts a multicenter, prospective, and observational cohort study design and does not involve randomization, control, and blinding. Patients with type 2 diabetes mellitus who were prescribed Dorzagliatin according to the package insert and physician's judgment in routine medical practice setting will be included, and the data of these patients during 52-week Dorzagliatin treatment will be collected to evaluate the safety of long-term medication.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must meet all of the following inclusion criteria to be eligible for this study:

1. Male or female ≥ 18 years of age at the time of signing the informed consent form;
2. Patients with type 2 diabetes mellitus diagnosed at screening;
3. Patients who have been prescribed Dorzagliatin according to the package insert and physician's judgment (the prescription should be made before enrolling the patient in this study and is independent of the enrollment decision);
4. Willingness to participate in the study and sign written informed consent.

Exclusion Criteria:

-

Patients will not be eligible if they meet any of the following criteria:

1. Other types of clinically diagnosed diabetes, such as type 1 diabetes or other special types of diabetes;
2. Patients who, in the opinion of the investigator, are at risk of allergy or intolerance to any component of Dorzagliatin;
3. Patients who, in the judgment of the investigator, cannot complete or are not suitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidences of ADRs and SAEs | 52 weeks
  The incidences of adverse drug reactions (ADRs) and serious adverse events (SAEs) as well as ADRs of special interest during the 52-week observation period of Dorzagliatin treatment.

SECONDARY OUTCOMES:
Blood glucose indicators | 52 weeks
  Changes from baseline in glycated hemoglobin (HbA1c), fasting plasma glucose (FPG), and 2-hour postprandial plasma glucose (2h-PPG) after 52 weeks of treatment with Dorzagliatin
Response rate | 52 weeks
  The proportion of patients with HbA1c < 7% after 52 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China